CLINICAL TRIAL: NCT03600883
Title: A Phase 1/2, Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Sotorasib (AMG 510) Monotherapy in Subjects With Advanced Solid Tumors With KRAS p.G12C Mutation and Sotorasib (AMG 510) Combination Therapy in Subjects With Advanced NSCLC With KRAS p.G12C Mutation (CodeBreaK 100)
Brief Title: A Phase 1/2, Study Evaluating the Safety, Tolerability, PK, and Efficacy of Sotorasib (AMG 510) in Subjects With Solid Tumors With a Specific KRAS Mutation (CodeBreaK 100)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20170543
Expanded Access: NCT04667234 (No longer available)
Record Dates: First submitted 2018-06-26; First posted 2018-07-26 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: KRAS p.G12C Mutant Advanced Solid Tumors
MeSH Terms: interventions — sotorasib; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1 Dose Exploration Part 1 monotherapy (Experimental): Cohorts with food effect and alternative dosing regimens
  Enrollment into the dose exploration cohorts may be from any eligible solid tumor type. Dose escalation will begin with 2-4 subjects treated at the lowest planned dose level of 180 mg. If no DLT is observed, dose escalation will continue to the next planned dose cohort
  Interventions: Drug: sotorasib
- Phase 1 Dose Expansion Part 2 monotherapy (Experimental): Upon completing the dose exploration part of the study, dose expansion may proceed with 3 groups consisting of subjects with KRAS p.G12C mutant advanced solid tumors. Dose expansion in these 3 groups may be done concurrently
  Interventions: Drug: sotorasib
- Phase 1 combination arm with sotorasib and anti PD-1/L1 (Experimental): Additional subjects will be enrolled into the combination arm with sotorasib in combination with an anti (PD-1/L1)
  Interventions: Drug: sotorasib; Drug: Anti PD-1/L1
- Phase 1 monotherapy treatment naive advanced NSCLC (Experimental): Separate cohort of part 1 dose expansion subjects to evaluate the safety and clinical activity of sotorasib administered orally once daily in subjects with previously untreated advanced non-small cell lung cancer (NSCLC). Drug-drug interaction will be evaluated in 6 of the subjects enrolled in the treatment naive cohort by adding Midazolam alone on Day -1 and in combination with sotorasib on Day 15 of Cycle 1, where each cycle is 21 days.
  Interventions: Drug: sotorasib; Drug: Midazolam
- Phase 2 monotherapy dose comparison (Experimental): Subjects with NSCLC will be enrolled in a dose comparison study evaluating safety and efficacy
  Interventions: Drug: sotorasib
- Phase 1 Does escalation and Expansion monotherapy BID (Experimental): BID 2L+solid tumors (fed state)
  Interventions: Drug: sotorasib

INTERVENTIONS:
Drug: sotorasib — Characterize the pharmacokinetics (PK) of sotorasib following administration as an oral Tablet formulation
Drug: Anti PD-1/L1 — Administered as an intravenous (IV) infusion
  Arms: Phase 1 combination arm with sotorasib and anti PD-1/L1
Drug: Midazolam — Administered as an oral hydrochloride (HCI) syrup
  Arms: Phase 1 monotherapy treatment naive advanced NSCLC

SUMMARY:
Evaluate the safety and tolerability of sotorasib in adult subjects with KRAS p.G12C mutant advanced solid tumors.

Estimate the maximum tolerated dose (MTD) and/or a recommended phase 2 dose (RP2D) in adult subjects with KRAS p.G12C mutant advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Men or women greater than or equal to 18 years old.
* Pathologically documented, locally-advanced or metastatic malignancy with, KRAS p.G12C mutation identified through molecular testing.

Exclusion Criteria

* Active brain metastases from non-brain tumors.
* Myocardial infarction within 6 months of study day 1.
* Gastrointestinal (GI) tract disease causing the inability to take oral medication.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 713 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary: Number of subjects with treatment-emergent adverse events | 24 Months
  Treatment-emergent adverse events will be a primary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 1 monotherapy treatment naïve advanced NSCLC
  * Phase 2 monotherapy dose comparison
Primary: Number of subjects with treatment-related adverse events | 24 Months
  Treatment-related adverse events will be a primary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 1 monotherapy treatment naïve advanced NSCLC
Primary: Number of subjects with grade ≥3 treatment-emergent adverse events | 24 Months
  Grade ≥3 treatment-emergent adverse events will be a primary outcome measure in the following group:
  - Phase 2 monotherapy dose comparison
Primary: Number of subjects with serious adverse events | 24 Months
  Serious adverse events will be a primary outcome measure in the following group:
  - Phase 2 monotherapy dose comparison
Primary: Number of subjects with adverse events of interest | 24 Months
  Adverse events of interest will be a primary outcome measure in the following group:
  - Phase 2 monotherapy dose comparison
Primary: Number of subjects with clinically significant changes in vital signs | Baseline to 24 Months
  Vital signs will be a primary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 1 monotherapy treatment naïve advanced NSCLC
Primary: Number of subjects with clinically significant changes in physical examination results | Baseline to 24 Months
  Physical examinations will be a primary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
Primary: Number of subjects with clinically significant changes on electrocardiograms (ECGs) | Baseline to 24 Months
  ECGs will be a primary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 1 monotherapy treatment naïve advanced NSCLC
Primary: Number of subjects with clinically significant changes in clinical laboratory values | Baseline to 24 Months
  Abnormal clinical laboratory values will be a primary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 1 monotherapy treatment naïve advanced NSCLC
Primary: Number of subjects with dose-limiting toxicities (DLTs) | 21 Days
  DLTs will be a primary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 1 monotherapy treatment naïve advanced NSCLC
Primary: Objective response rate (ORR) as assessed by RECIST 1.1 criteria | 24 Months
  ORR will be a primary outcome measure in the following group:
  * Phase 1 monotherapy treatment naïve advanced NSCLC
  * Phase 2 monotherapy
  * Phase 2 monotherapy dose comparison
Primary: Duration of response (DOR) as assessed by RECIST 1.1 criteria | 24 Months
  DOR will be a primary outcome measure in the following group:
  - Phase 1 monotherapy treatment naïve advanced NSCLC
Primary: Disease control as assessed by RECIST 1.1 criteria | 24 Months
  Disease control will be a primary outcome measure in the following group:
  - Phase 1 monotherapy treatment naïve advanced NSCLC
Primary: Duration of stable disease (SD) as assessed by RECIST 1.1 criteria | 24 Months
  Duration of SD will be a primary outcome measure in the following group:
  - Phase 1 monotherapy treatment naïve advanced NSCLC
Primary: Time to response (TTR) as assessed by RECIST 1.1 criteria | 24 Months
  TTR will be a primary outcome measure in the following group:
  - Phase 1 monotherapy treatment naïve advanced NSCLC

SECONDARY OUTCOMES:
Secondary: Plasma concentration (Cmax) of sotorasib | 15 Weeks
  Cmax will be a secondary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 1 monotherapy treatment naïve advanced NSCLC
  * Phase 2 monotherapy dose comparison
Secondary: Plasma concentration (Cmax) of midazolam | 16 Days
  Cmax of midazolam will be a secondary outcome measure for the subgroup of subjects who were administered midazolam in the following group:
  - Phase 1 monotherapy treatment naïve advanced NSCLC
Secondary: Time to achieve Cmax (Tmax) of sotorasib | 15 Weeks
  Tmax will be a secondary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 1 monotherapy treatment naïve advanced NSCLC
Secondary: Area under the plasma concentration-time curve (AUC) of sotorasib | 15 Weeks
  AUC will be a secondary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 1 monotherapy treatment naïve advanced NSCLC
  * Phase 2 monotherapy dose comparison
Secondary: Area under the plasma concentration-time curve (AUC) of midazolam | 16 Days
  AUC of midazolam will be a secondary outcome measure for the subgroup of subjects who were administered midazolam in the following group:
  - Phase 1 monotherapy treatment naïve advanced NSCLC
Secondary: Clearance of midazolam from the plasma | 16 Days
  Clearance of midazolam from the plasma will be a secondary outcome measure for the subgroup of subjects who were administered midazolam in the following group:
  - Phase 1 monotherapy treatment naïve advanced NSCLC
Secondary: Terminal half-life (t1/2) of midazolam | 16 Days
  t1/2 of midazolam will be a secondary outcome measure for the subgroup of subjects who were administered midazolam in the following group:
  - Phase 1 monotherapy treatment naïve advanced NSCLC
Secondary: Objective response rate (ORR) as assessed by RECIST 1.1 criteria | 24 Months
  ORR will be a secondary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
Secondary: Duration of response (DOR) as assessed by RECIST 1.1 criteria | 24 Months
  DOR will be a secondary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 2 monotherapy dose comparison
Secondary: Disease control as assessed by RECIST 1.1 criteria | 24 Months
  DOR will be a secondary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 2 monotherapy dose comparison
Secondary: Progression-free survival (PFS) as assessed by RECIST 1.1 criteria | 24 Months
  PFS will be a secondary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 2 monotherapy dose comparison
  * Phase 1 monotherapy treatment naïve advanced NSCLC
Secondary: Duration of stable disease (SD) as assessed by RECIST 1.1 criteria | 24 Months
  Duration of SD will be a secondary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
Secondary: Depth of response (best percentage change from baseline in lesion sum diameters) as assessed by RECIST 1.1 criteria | Baseline to 24 Months
  Depth of response will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy dose comparison
Secondary: Time to response (TTR) as assessed by RECIST 1.1 criteria | 24 Months
  DOR will be a secondary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 2 monotherapy dose comparison
Secondary: Overall survival (OS) | 24 Months
  OS will be a secondary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
  * Phase 2 monotherapy
  * Phase 1 combination arm with sotorasib and anti PD-1/L1
  * Phase 2 monotherapy dose comparison
  * Phase 1 monotherapy treatment naïve advanced NSCLC
Secondary: sotorasib exposure and QTc interval relationship | 24 Months
  sotorasib exposure and QTc interval relationship will be a secondary outcome measure for the following groups:
  * Phase 1 Dose Exploration Part 1 monotherapy
  * Phase 1 Dose Expansion Part 2 monotherapy
Secondary: Progression-free survival (PFS) at 6 months | 6 Months
  PFS at 6 months will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy
Secondary: Progression-free survival (PFS) at 12 months | 12 Months
  PFS at 12 months will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy
Secondary: Overall survival (OS) at 12 months | 12 Months
  OS at 12 months will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy
Secondary: Number of subjects with treatment-emergent adverse events | 24 Months
  Treatment-emergent adverse events will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy
Secondary: Number of subjects with grade ≥3 treatment-emergent adverse events | 24 Months
  Grade ≥3 treatment-emergent adverse events will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy
Secondary: Impact of treatment on disease-related symptoms and health related quality of life (HRQOL) as assessed by EORTC QLQ-C30 | 24 Months
  Impact of treatment on disease-related symptoms and HRQOL will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy dose comparison
Secondary: Impact of treatment on disease-related symptoms and HRQOL as assessed by disease-specific modules Quality-of-Life Questionnaire Lung Cancer Module (QLQ LC13) | 24 Months
  Impact of treatment on disease-related symptoms and HRQOL will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy dose comparison
Secondary: Impact of treatment on disease-related symptoms and HRQOL as assessed by non-small cell lung cancer symptom assessment questionnaire (NSCLC SAQ) for NSCLC | 24 Months
  Impact of treatment on disease-related symptoms and HRQOL will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy dose comparison
Secondary: Impact of treatment on disease-related symptoms and HRQOL as assessed by Patient Global Impression of Severity (PGIS) | 24 Months
  Impact of treatment on disease-related symptoms and HRQOL will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy dose comparison
Secondary: Impact of treatment on disease-related symptoms and HRQOL as assessed by Patient Global Impression of Change (PGIC) in cough, dyspnea and chest pain for NSCLC | 24 Months
  Impact of treatment on disease-related symptoms and HRQOL will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy dose comparison
Secondary: Treatment-related symptoms and impact on the subject as assessed by EORTC QLQ-C30 | 24 Months
  Treament related symptoms and impact on the subject will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy dose comparison
Secondary: Treatment-related symptoms and impact on the subject as assessed by selected questions from the Patient-reported Outcome of the Common Terminology Criteria for Adverse Events (PRO-CTCAE library) | 24 Months
  Treatment-related symptoms and impact on the subject will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy dose comparison
Secondary: Treatment-related symptoms and impact on the subject as assessed by a single item about symptom bother, item GP5 of the Functional Assessment of Cancer Therapy - General (FACT-G) | 24 Months
  Treatment-related symptoms and impact on the subject will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy dose comparison
Secondary: Change from baseline in physical function as assessed by EORTC QLQ-C30 | Baseline to 24 Months
  Treatment-related symptoms and impact on the subject will be a secondary outcome measure for the following group:
  - Phase 2 monotherapy dose comparison

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (133):
- United States (39):
  - City of Hope National Medical Center, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - University of California at SF, San Francisco, California
  - Sarcoma Oncology Research Center LLC, Santa Monica, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Medical Oncology Hematology Consultants Helen F Graham Cancer Center, Newark, Delaware
  - University of Florida Health, Gainesville, Florida
  - AdventHealth Orlando Infusion Center, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at New York University Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Morris Cancer Clinic, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Cancer Pavillion, Pittsburgh, Pennsylvania
  - Gibbs Cancer Center and Research Institute - Spartanburg, Spartanburg, South Carolina
  - Vanderbilt University Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology - Austin Central, Austin, Texas
  - Texas Oncology - Baylor, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - US Oncology Research Investigational Products Center, Fairfax, Virginia
  - Virginia Cancer Specialists PC, Fairfax, Virginia
  - Blue Ridge Cancer Care, Salem, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (4):
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Peter MacCallum Cancer Centre, Parkville, Victoria
- Austria (5):
  - Medizinische Universitaet Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Universitaetsklinikum Krems, Krems
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf, Vienna
- Belgium (9):
  - Institut Jules Bordet, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege, Liège
  - AZ Delta Campus Rumbeke, Roeselare
- Brazil (6):
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Nucleo de Novos Tratamentos em Cancer, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo, São Paulo
  - Oncologia Rede D´Or, São Paulo, São Paulo
  - Instituto Coi, Rio de Janeiro
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - London Regional Cancer Program, London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre Glen Site, Montreal, Quebec
- France (6):
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hopital de la Timone, Marseille
  - Institut Curie, Paris
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Germany (3):
  - Universitatsklinikum Koln, Cologne
  - Universitätsklinikum Essen, Essen
  - Klinikum der Universität München Campus Grosshadern, München
- Greece (5):
  - Henry Dunant Hospital Center, Athens
  - Metropolitan Hospital, Athens
  - University Hospital of Heraklion, Heraklion - Crete
  - Theagenion Cancer Hospital, Thessaloniki
  - Agios Loukas Clinic, Thessaloniki
- Hungary (6):
  - Semmelweis Egyetem, Budapest
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Szent Borbala Korhaz, Tatabánya
  - Tudogyogyintezet Torokbalint, Törökbálint
- Japan (15):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - St Marianna University Hospital, Kawasaki-shi, Kanagawa
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Portugal (5):
  - Fundacao Champalimaud, Lisbon
  - Centro Hospitalar Universitario de Lisboa Norte EPE - Hospital Pulido Valente, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Centro Hospitalar Universitario do Porto EPE - Hospital de Santo Antonio, Porto
  - Hospital Cuf porto, Porto
- Romania (8):
  - Institutul Oncologic, Prof Dr Alexandru Trestioreanu, Bucharest
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - SC Medisprof SRL, Cluj-Napoca
  - Centrul de Radioterapie Amethyst Cluj, Cluj-Napoca
  - Centrul de Oncologie Sf Nectarie SRL, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Municipal Ploiesti, Ploieşti
  - SC Oncomed SRL, Timișoara
- South Korea (7):
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Clinica Universidad de Navarra, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
- Switzerland (3):
  - Universitaetsspital Basel, Basel
  - Hopitaux Universitaires de Geneve, Geneva
  - Universitaetsspital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Canon J, Rex K, Saiki AY, Mohr C, Cooke K, Bagal D, Gaida K, Holt T, Knutson CG, Koppada N, Lanman BA, Werner J, Rapaport AS, San Miguel T, Ortiz R, Osgood T, Sun JR, Zhu X, McCarter JD, Volak LP, Houk BE, Fakih MG, O'Neil BH, Price TJ, Falchook GS, Desai J, Kuo J, Govindan R, Hong DS, Ouyang W, Henary H, Arvedson T, Cee VJ, Lipford JR. The clinical KRAS(G12C) inhibitor AMG 510 drives anti-tumour immunity. Nature. 2019 Nov;575(7781):217-223. doi: 10.1038/s41586-019-1694-1. Epub 2019 Oct 30. PMID 31666701
- [Background] Skoulidis F, Li BT, Dy GK, Price TJ, Falchook GS, Wolf J, Italiano A, Schuler M, Borghaei H, Barlesi F, Kato T, Curioni-Fontecedro A, Sacher A, Spira A, Ramalingam SS, Takahashi T, Besse B, Anderson A, Ang A, Tran Q, Mather O, Henary H, Ngarmchamnanrith G, Friberg G, Velcheti V, Govindan R. Sotorasib for Lung Cancers with KRAS p.G12C Mutation. N Engl J Med. 2021 Jun 24;384(25):2371-2381. doi: 10.1056/NEJMoa2103695. Epub 2021 Jun 4. PMID 34096690
- [Background] Fakih MG, Kopetz S, Kuboki Y, Kim TW, Munster PN, Krauss JC, Falchook GS, Han SW, Heinemann V, Muro K, Strickler JH, Hong DS, Denlinger CS, Girotto G, Lee MA, Henary H, Tran Q, Park JK, Ngarmchamnanrith G, Prenen H, Price TJ. Sotorasib for previously treated colorectal cancers with KRASG12C mutation (CodeBreaK100): a prespecified analysis of a single-arm, phase 2 trial. Lancet Oncol. 2022 Jan;23(1):115-124. doi: 10.1016/S1470-2045(21)00605-7. Epub 2021 Dec 15. PMID 34919824
- [Background] Hong DS, Fakih MG, Strickler JH, Desai J, Durm GA, Shapiro GI, Falchook GS, Price TJ, Sacher A, Denlinger CS, Bang YJ, Dy GK, Krauss JC, Kuboki Y, Kuo JC, Coveler AL, Park K, Kim TW, Barlesi F, Munster PN, Ramalingam SS, Burns TF, Meric-Bernstam F, Henary H, Ngang J, Ngarmchamnanrith G, Kim J, Houk BE, Canon J, Lipford JR, Friberg G, Lito P, Govindan R, Li BT. KRASG12C Inhibition with Sotorasib in Advanced Solid Tumors. N Engl J Med. 2020 Sep 24;383(13):1207-1217. doi: 10.1056/NEJMoa1917239. Epub 2020 Sep 20. PMID 32955176
- [Background] Zhao Y, Murciano-Goroff YR, Xue JY, Ang A, Lucas J, Mai TT, Da Cruz Paula AF, Saiki AY, Mohn D, Achanta P, Sisk AE, Arora KS, Roy RS, Kim D, Li C, Lim LP, Li M, Bahr A, Loomis BR, de Stanchina E, Reis-Filho JS, Weigelt B, Berger M, Riely G, Arbour KC, Lipford JR, Li BT, Lito P. Diverse alterations associated with resistance to KRAS(G12C) inhibition. Nature. 2021 Nov;599(7886):679-683. doi: 10.1038/s41586-021-04065-2. Epub 2021 Nov 10. PMID 34759319
- [Background] Dy GK, Govindan R, Velcheti V, Falchook GS, Italiano A, Wolf J, Sacher AG, Takahashi T, Ramalingam SS, Dooms C, Kim DW, Addeo A, Desai J, Schuler M, Tomasini P, Hong DS, Lito P, Tran Q, Jones S, Anderson A, Hindoyan A, Snyder W, Skoulidis F, Li BT. Long-Term Outcomes and Molecular Correlates of Sotorasib Efficacy in Patients With Pretreated KRAS G12C-Mutated Non-Small-Cell Lung Cancer: 2-Year Analysis of CodeBreaK 100. J Clin Oncol. 2023 Jun 20;41(18):3311-3317. doi: 10.1200/JCO.22.02524. Epub 2023 Apr 25. PMID 37098232
- [Background] Dy GK, Govindan R, Velcheti V, Falchook GS, Italiano A, Wolf J, Sacher AG, Takahashi T, Ramalingam SS, Dooms C, Kim DW, Addeo A, Desai J, Schuler M, Tomasini P, Hong DS, Lito P, Tran Q, Jones S, Anderson A, Hindoyan A, Snyder W, Skoulidis F, Li BT. Long-term benefit of sotorasib in patients with KRAS G12C-mutated non-small-cell lung cancer: plain language summary. Future Oncol. 2024 Jan;20(3):113-120. doi: 10.2217/fon-2023-0560. Epub 2023 Nov 27. PMID 38010044
- [Background] Dilly J, Hoffman MT, Abbassi L, Li Z, Paradiso F, Parent BD, Hennessey CJ, Jordan AC, Morgado M, Dasgupta S, Uribe GA, Yang A, Kapner KS, Hambitzer FP, Qiang L, Feng H, Geisberg J, Wang J, Evans KE, Lyu H, Schalck A, Feng N, Lopez AM, Bristow CA, Kim MP, Rajapakshe KI, Bahrambeigi V, Roth JA, Garg K, Guerrero PA, Stanger BZ, Cristea S, Lowe SW, Baslan T, Van Allen EM, Mancias JD, Chan E, Anderson A, Katlinskaya YV, Shalek AK, Hong DS, Pant S, Hallin J, Anderes K, Olson P, Heffernan TP, Chugh S, Christensen JG, Maitra A, Wolpin BM, Raghavan S, Nowak JA, Winter PS, Dougan SK, Aguirre AJ. Mechanisms of Resistance to Oncogenic KRAS Inhibition in Pancreatic Cancer. Cancer Discov. 2024 Nov 1;14(11):2135-2161. doi: 10.1158/2159-8290.CD-24-0177. PMID 38975874
- [Background] Hochmair MJ, Vermaelen K, Mountzios G, Carcereny E, Dooms C, Lee SH, Morocz E, Kato T, Ciuleanu TE, Dy GK, Parente B, O'Byrne KJ, Chu QS, Castro Junior G, Girard N, Snyder W, Tran Q, Kormany W, Houk B, Mehta B, Curioni-Fontecedro A. Sotorasib (960 mg or 240 mg) once daily in patients with previously treated KRAS G12C-mutated advanced NSCLC. Eur J Cancer. 2024 Sep;208:114204. doi: 10.1016/j.ejca.2024.114204. Epub 2024 Jul 5. PMID 39029295
- [Background] Nagase M, Houk B, Vuu I, Cardona P, Dutta S, Lin CW. Population Pharmacokinetics of Sotorasib in Healthy Subjects and Advanced Solid Tumor Patients Harboring a KRASG12C Mutation from Phase 1 and Phase 2 Studies. AAPS J. 2025 Jan 13;27(1):26. doi: 10.1208/s12248-024-01013-6. PMID 39806205
- [Derived] Strickler JH, Satake H, George TJ, Yaeger R, Hollebecque A, Garrido-Laguna I, Schuler M, Burns TF, Coveler AL, Falchook GS, Vincent M, Sunakawa Y, Dahan L, Bajor D, Rha SY, Lemech C, Juric D, Rehn M, Ngarmchamnanrith G, Jafarinasabian P, Tran Q, Hong DS. Sotorasib in KRAS p.G12C-Mutated Advanced Pancreatic Cancer. N Engl J Med. 2023 Jan 5;388(1):33-43. doi: 10.1056/NEJMoa2208470. Epub 2022 Dec 21. PMID 36546651
- [Derived] Lanman BA, Allen JR, Allen JG, Amegadzie AK, Ashton KS, Booker SK, Chen JJ, Chen N, Frohn MJ, Goodman G, Kopecky DJ, Liu L, Lopez P, Low JD, Ma V, Minatti AE, Nguyen TT, Nishimura N, Pickrell AJ, Reed AB, Shin Y, Siegmund AC, Tamayo NA, Tegley CM, Walton MC, Wang HL, Wurz RP, Xue M, Yang KC, Achanta P, Bartberger MD, Canon J, Hollis LS, McCarter JD, Mohr C, Rex K, Saiki AY, San Miguel T, Volak LP, Wang KH, Whittington DA, Zech SG, Lipford JR, Cee VJ. Discovery of a Covalent Inhibitor of KRASG12C (AMG 510) for the Treatment of Solid Tumors. J Med Chem. 2020 Jan 9;63(1):52-65. doi: 10.1021/acs.jmedchem.9b01180. Epub 2019 Dec 24. PMID 31820981
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com